CLINICAL TRIAL: NCT02220179
Title: Resilience for Children and Young People
Brief Title: Resilience for Children and Young People in Foster Care and Residential Care in Denmark
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Poul Bak (Other)
Collaborators: TRYG Foundation (Other)
Responsible Party: Sponsor-Investigator, Poul Bak, MD, University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: DK-res-care
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Children and Adolescents in Foster Care and Residential Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (No Intervention): service as usual
- Intervention group 1 (Experimental): Participants are offered access to the web based resilience program
  Interventions: Behavioral: The Resilience Program
- Intervention group 2 (Experimental): Participants are offered access to the web based resilience program and are also invited to join a short introduction course about the program
  Interventions: Behavioral: The Resilience Program

INTERVENTIONS:
Behavioral: The Resilience Program — Se the CONSORT trial protocol at http://myresilience.org/ at the subsite 'about us'
  Arms: Intervention group 1; Intervention group 2

SUMMARY:
In this project we invite 9.000 children and young persons in Denmark and their foster parents and staff at the residential institutions to participate in a cluster randomized controlled intervention study where we aim to test the effectiveness of a web based knowledge and inspiration program about resilience for children, adolescents and adults (called myresilience.org). The complete CONSORT trial protocol is available at http://myresilience.org/ at the subsite 'about us'.

DETAILED DESCRIPTION:
The complete CONSORT trial protocol is available at http://myresilience.org/ at the subsite 'about us'.

ELIGIBILITY:
Inclusion Criteria:

* All children and adolescents registered in foster care in Denmark on august 11th 2014.
* All children and adolescents registered in residential care in Denmark on august 11th 2014.

Exclusion Criteria:

• Request for legal protection against contacts from researchers.

Max Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9000 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
National Test in Danish Reading | Outcome data will be collected on the average 2 years after intervention
  The National test in danish reading is a standard performance test which is mandatory for all danish student. It is administered for every other year.

SECONDARY OUTCOMES:
The frequency of Care collapse | Outcome data will be collected on the average 2 years after intervention
  All incidents of collapse in a care relation is registered by the danish authorities. The informations in this register are used for this outcome measure.

OTHER OUTCOMES:
Questionnaire data | data collected august 2015
  Se the trial CONSORT protocol at http://myresilience.org/ at the subsite 'about us'

CONTACTS AND LOCATIONS:
Overall Officials: Poul L Bak, MD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark, Denmark

REFERENCES:
- See also: Find the CONSORT trial protocol on the subsite 'about us' — http://myresilience.org/